CLINICAL TRIAL: NCT04645862
Title: Prospective 4D CTA of BAV Competence
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 843190
Record Dates: First submitted 2020-11-13; First posted 2020-11-27 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Bicuspid
Keywords: bicuspid aortic valve
MeSH Terms: conditions — Bicuspid Aortic Valve Disease | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CT scans — 4D CTA imaging

SUMMARY:
The study involves annual 4D CTA imaging of the bicuspid aortic valve for a period of 5 years. CTA is often standard of care for BAV patients, but patients in this study will receive a higher radiation dose with a 4D imaging protocol. There may also be patients enrolled in the study who have a 4D CTA for research purposes when a routine CTA is not required for clinical care.

DETAILED DESCRIPTION:
The bicuspid aortic valve (BAV) is the most common congenital heart disease. The purpose of this study is to better understand the anatomy of physiologically normal, or competent, BAVs without stenosis or insufficiency (AI) in order to support evidence-based standardization of BAV repair surgery. Men and women over 18 years of age with a diagnosis of BAV and minimal aortic valve calcification at baseline will undergo annual 4D computed tomography angiography (CTA) scans, routine transthoracic echocardiograms, and history and physical assessments over the course of the 5-year study period. Patients who are pregnant, have renal insufficiency (creatinine 2 mg/dL), or who have a contraindication to intravenous contrast will be excluded. Patients will be stratified into study groups according to baseline AI: approximately half of patients will have no to mild AI at baseline and the other half will have moderate to severe AI at baseline. Anatomical measurements will be obtained from the 4D CTA scans and analyzed at each phase of the cardiac cycle, as well as longitudinally. The 4D CTA imaging and analysis will not impact medical care of the study participants; the anatomical measurements will be used in the future as evidence-based standards for determining valve repair candidacy for BAV patients with AI.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Documented bicuspid aortic valve identified via clinical imaging (e.g., CT, MRI, or echocardiogram) with minimal calcification at the time of enrollment
* Participant must sign the informed consent form

Exclusion Criteria:

* Pregnancy (determined by point of care urine pregnancy test)
* Renal failure (estimated Glomerular Filtration Rate (eGFR) < 30), precluding them from receiving intravenous contrast)
* Documentation of previous intravenous contrast allergy (unless they are having a CT with steroid preparation as part of routine clinical care)
* Previous aortic valve replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bicuspid aortic valve identified via clinical imaging
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cusp surface areas over the cardiac cycle | Through study completion, an average of 1 year
  Surface area of each cusp in mm2 in one cardiac cycle (~0.6 - 1s in length). This measurement is made directly from the CT image.
Cusp height (geometric and effective) | Through study completion, an average of 1 year
  Geometric and effective cusp height in mm in one cardiac cycle (~0.6 - 1s in length). This measurement is made directly from the CT image.
Cusp free margin length | Through study completion, an average of 1 year
  Length of the free margin of each cusp in mm in one cardiac cycle (~0.6 - 1s in length). This measurement is made directly from the CT image.
Cusp thickness (including raphe thickness, if applicable) | Through study completion, an average of 1 year
  Thickness of each cusp in mm in one cardiac cycle (~0.6 - 1s in length). This measurement is made directly from the CT image.
Commissural height | Through study completion, an average of 1 year
  Height of each commissure in mm in one cardiac cycle (~0.6 - 1s in length). This measurement is made directly from the CT image.
Sino tubular junction size | Through study completion, an average of 1 year
  Diameter of the sinotubular junction in mm in one cardiac cycle (~0.6 - 1s in length). This measurement is made directly from the CT image.
Size of the sinuses of Valsalva | Through study completion, an average of 1 year
  Maximum diameter of the sinuses of Valsalva (mid-level of the aortic root) in mm in one cardiac cycle (~0.6 - 1s in length). This measurement is made directly from the CT image.
Ventriculoaortic junction size | Through study completion, an average of 1 year
  Diameter of the ventriculoaortic junction in mm in one cardiac cycle (~0.6 - 1s in length). This measurement is made directly from the CT image.
Aortic annulus size | Through study completion, an average of 1 year
  Diameter of the aortic cusp in mm measured in one cardiac cycle (~0.6 - 1s in length). This measurement is made directly from the CT image.
Coaptation height at diastole | Through study completion, an average of 1 year
  Length of the coaptation zone of the cusps in mm when the valve is closed. This measurement is made in one cardiac cycle (~0.6 - 1s in length) from the CT image.
Cusp displacement over the cardiac cycle | Through study completion, an average of 1 year
  Total displacement of the center of the free margin of each cusp in mm during one cardiac cycle (~0.6 - 1s in length). This measurement is made directly from the CT image.
Cusp velocity over the cardiac cycle | Through study completion, an average of 1 year
  Maximum velocity of the center of the free margin of each cusp in mm/s during one cardiac cycle (~0.6 - 1s in length). This measurement is made directly from the CT image.
Size of the ascending aorta | Through study completion, an average of 1 year
  Maximum diameter of the ascending aorta in cm during one cardiac cycle (~0.6 - 1s in length). This measurement is made directly from the CT image.

SECONDARY OUTCOMES:
Development of aortic insufficiency and/or stenosis. | Through study completion, an average of 1 year
  Degree of aortic insufficiency as measured on standard-of-care echocardiography
Development of aortic insufficiency and/or stenosis. | Through study completion, an average of 1 year
  The need for surgical intervention for disease of the aortic valve and/or ascending aorta

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT04645862/Prot_000.pdf